CLINICAL TRIAL: NCT03207724
Title: A Phase I Study of Onivyde and 5-FU in Combination With Xilonix for Advanced Pancreatic Cancer With Cachexia
Brief Title: Study of Onivyde and 5-FU in Combination With Xilonix for Pancreatic Cancer With Cachexia
Acronym: OnFX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Andrew Hendifar, MD (Other)
Collaborators: Ipsen (Industry); Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor-Investigator, Andrew Hendifar, MD, Assistant Professor of Medicine, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2016-07-Hendifar-OnFX
Record Dates: First submitted 2017-06-30; First posted 2017-07-05 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Pancreatic Cancer; Cachexia; Weight Loss
Keywords: advanced pancreatic cancer; locally advanced pancreatic cancer; recurrent diagnosis; new diagnosis; adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms; Cachexia; Weight Loss; Disease; Adenocarcinoma | interventions — bermekimab; irinotecan sucrosofate; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Xilonix plus Onivyde and 5FU (Experimental): interleukin-1-alpha antagonist (Xilonix) in addition to standard chemotherapy of onivyde and 5-fluorouracil/folinic acid (leucovorin)
  Interventions: Drug: Xilonix plus Onivyde and 5FU

INTERVENTIONS:
Drug: Xilonix plus Onivyde and 5FU — Xilonix by IV
  Other Names: interleukin-1-alpha antagonist

SUMMARY:
This study is being conducted to examine the safety of the investigational drug, Xilonix(™), in addition to standard doses of Onivyde® (nanoliposomal irinotecan) and 5- fluorouracil (5FU)/folinic acid (leucovorin) for pancreatic cancer patients with cachexia. Cachexia is a syndrome that includes involuntary weight loss and physical deterioration that can contribute to poor outcomes of cancer treatment. In other studies, Xilonix has increased lean body mass in advanced cancer patients. This increase could lead to improved weight maintenance and quality of life.

DETAILED DESCRIPTION:
This study will prospectively evaluate advanced pancreatic adenocarcinoma patients. The intervention will be interleukin-1-alpha antagonist (Xilonix) in addition to standard chemotherapy. The first aim is to assess the safety and identify the maximum tolerated dose of Onivyde with 5-fluorouracil/folinic acid in combination with the study agent, Xilonix. The study will also create a repository of serum, tissue, and fecal specimens to investigate novel biomarkers related to cachexia with pancreatic adenocarcinoma and interleukin-1-alpha blockade. Lastly, the study will assess for a correlation between cachexia, activity, and PROs on domains of quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or locally advanced pancreatic cancer patients (can include new or recurrent diagnosis) referred to SOCCI-CSMC for chemotherapy that has progressed through or intolerant to gemcitabine based chemotherapy
* Cachexia defined as greater than 5% unexplained weight loss within any 6 month period prior to screening visit OR as documented by the medical physician based on standard diagnosis of cachexia
* Age ≥ 18 years
* ECOG performance status 0-2 or Karnofsky PS >60%
* Patients must have normal organ and marrow function
* Ability to understand and the willingness to sign a written informed consent
* Negative pregnancy test for WOCBP
* WOCBP and men must agree to use of adequate contraception

Exclusion Criteria:

* Patients who are currently receiving any other investigational agents
* Patients who have received more than one chemotherapeutic regimen in metastatic setting
* Patients with CNS metastases
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with unresolved grade 3/4 adverse effects of prior therapy at time of enrollment
* Subjects with history of hypersensitivity to compounds of similar chemical or biologic composition to Xilonix or Onivyde
* Women who are pregnant or breastfeeding
* Dementia or altered mental status that would prohibit the understanding or rendering of informed consent
* Patients with known Dihydropyrimidine dehydrogenase deficiency (DPD deficiency)
* Patients known to be UGT1A1*28 allele homozygous
* Patients who have had a live vaccine within 3 months of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2020-10-27 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Dose Limiting Toxicities (DLT) in the First Cycle for the determination of the Maximum Tolerated Dose (MTD) | 28 days (first cycle)
  Assess safety of novel combination
Maximum Tolerated Dose (MTD) of onivyde, 5-fluorouracil/folinic acid in combination with Xilonix | 28 days (first cycle)
  Assess MTD of Onivyde in combination with novel therapy

SECONDARY OUTCOMES:
Weight stability | 6 months
  Mean change from baseline (kg) up to 6 months
Lean Body Mass | 6 months
  Mean change from baseline (kg) up to 6 months
Overall Survival | 12 months
  To measure overall survival up to 12 months from baseline
Progression Free Survival | 12 months
  To measure progression free survival up to 12 months from baseline
Mean change in global quality of life (QOL) score (EORTC Pan26) | 6 months
  Assessment based on patient-reported QOL up to 6 months from baseline
Mean change in global score of patient-reported response to therapy (FAACT questionnaire- Functional Assessment of Anorexia/Cachexia Therapy) | 6 months
  Assessment based on patient-reported outcomes up to 6 months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Hendifar, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gong J, Thomassian S, Kim S, Gresham G, Moshayedi N, Ye JY, Yang JC, Jacobs JP, Lo S, Nissen N, Gaddam S, Tighiouart M, Osipov A, Hendifar A. Phase I trial of Bermekimab with nanoliposomal irinotecan and 5-fluorouracil/folinic acid in advanced pancreatic ductal adenocarcinoma. Sci Rep. 2022 Sep 2;12(1):15013. doi: 10.1038/s41598-022-19401-3. PMID 36056179